CLINICAL TRIAL: NCT05569174
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter, 24-week Study Investigating the Efficacy and Safety of Secukinumab Compared to Placebo in Adult Patients With Moderate to Severe Rotator Cuff Tendinopathy and Failure to Conventional Therapy
Brief Title: Study of Efficacy and Safety of AIN457/Secukinumab in Patients With Rotator Cuff Tendinopathy
Acronym: UnchAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457FDE05; 2022-001516-26 (EudraCT Number)
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Tendinopathy
Keywords: shoulder; rotator cuff; IL-17A-Ab; AIN457X; Impingement syndrome
MeSH Terms: conditions — Tendinopathy | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Participants received 300 mg of secukinumab s.c. for 12 weeks
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Participants received placebo s.c. for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 300 mg s.c for 12 weeks in a pre-filled syringe (PFS)
  Other Names: AIN457
  Arms: Secukinumab
Other: Placebo — Placebo to match secukinumab s.c. for 12 weeks in a PFS
  Arms: Placebo

SUMMARY:
The purpose of this study was to investigate the efficacy and safety of secukinumab subcutaneously (s.c.) compared to placebo in adult patients with moderate to severe rotator cuff tendinopathy and failure to conventional therapy.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, parallel-group, multicenter, Phase IIIb, 24-week study to investigate the superior efficacy of secukinumab and safety in participants with rotator cuff tendinopathy.

Secukinumab 300 mg s.c. was compared to placebo (both arms in combination with patient individualized conventional therapy) in relieving clinical symptoms at Week 24.

The study consisted of a screening period up to 6 weeks, a 2-week run-in period, a 12-week treatment period and a 12-week follow-up period. Treatment and follow-up periods were blinded. Participants who met the eligibility criteria at screening continued to the run-in period and were randomized. In the run-in period, participants performed 2 weeks of home-based standardized physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent had to be obtained prior to participation in the study.
* Males and non-pregnant, non-nursing females were between 18 and 65 years of age.
* Rotator cuff tendinopathy (unilateral) was present with a positive "Painful Arc Test" on examination.
* Symptoms had been present for at least 6 weeks but not more than 6 months at Baseline.
* Moderate to severe rotator cuff tendinopathy was demonstrated by all of the following criteria:

  1. WORC score was ≤ 40 at Baseline.
  2. NRS pain score was ≥ 5 at Baseline and for at least 3 days of the 7 days prior to Baseline.
  3. Nocturnal pain occurred at least 4 out of the 7 days in the week prior to Baseline.
* Patients had failed at least 8 weeks of conventional therapy prior to Baseline: inadequate response to NSAIDs and/or paracetamol and physiotherapy; or intolerance to NSAIDs and/or paracetamol.

Exclusion Criteria:

* Greater than 50% partial thickness tear had been established by MRI or ultrasound during assessment in the Run-in phase.
* Patients were expected to require glucocorticoid treatment throughout the trial duration at Baseline (e.g., systemic, intramuscular, local injections in shoulder).
* Previous surgery, or plans for surgery, during the study period, in the affected shoulder.
* Rheumatologic and chronic inflammatory diseases, including but not limited to inflammatory bowel disease, polymyalgia rheumatica (PMR), PsA, axSpA and rheumatoid arthritis (RA), fibromyalgia or - severe pain disorder unrelated to the target shoulder.
* Rheumatoid factor (RF) and anti-cyclic citrullinated peptide (anti-CCP) antibodies were positive at Screening.
* History of adhesive capsulitis/frozen shoulder or calcification in the tendon (in affected or contralateral shoulder) had been confirmed clinically or by medical imaging.
* Symptomatic osteoarthritis of the shoulder (glenohumeral, acromioclavicular) in affected or contralateral shoulder had been confirmed by medical imaging.
* Patients had traumatic rupture that would have been considered eligible for surgery for repair of cuff tear.
* Neurological conditions including but not limited to cervical radiculopathy, which in the opinion of the investigator could have explained the patient's symptoms.
* Any intra-articular/subacromial glucocorticoid treatment had occurred within 12 weeks prior to Baseline or more than 2 injections for the current tendinopathy.
* Any oral, intramuscular or i.v. glucocorticoid treatment had occurred 12 weeks prior to Baseline or during the current tendinopathy, whichever was longer.
* Previous platelet rich plasma (PRP) injections or fluoroquinolone/quinolone antibiotics had occurred within 12 weeks prior to Baseline or during the current tendinopathy, whichever was longer.
* Neuromuscular or primary/secondary muscular deficiency had limited the ability to perform functional measurement (e.g., shoulder strength test).
* Previous hyaluronic injections had occurred within 12 weeks prior to Baseline or during the current tendinopathy, whichever was longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- Germany (16):
  - Novartis Investigative Site, Karlsruhe, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Gladbeck
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heinsberg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Schönebeck

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=3085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized in 19 study sites across Germany
Pre-assignment Details: A total of 100 participants were screened and 62 participants were randomized in nearly equal numbers to the 2 treatment groups (secukinumab: N=30; placebo: N=32) and received study treatment
Period: Overall Study
Arm/Group | Secukinumab | Placebo
Started | 30 | 32
Completed | 30 | 27
Not Completed | 0 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Lack of compliance | 0 | 1
Not completed — Withdrawal of consent | 0 | 1
Not completed — Participant wish | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (7.5) | 52.1 (9.0) | 52.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 10 | 17 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 29 | 31 | 60
  Black | 1 | 0 | 1
  Asian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Western Ontario Rotator Cuff (WORC) Patient Reported Outcome (PRO) Percentage Score at Week 24
Description: The WORC Index consisted of 21 items divided into 5 Domains: Physical Symptoms (6 items), Sport/Recreation (4 items), Work Function (4 items), Lifestyle Function (4 items) and Emotional Function (3 items). Each of the 21 items in the WORC was rated using a visual analogue scale (VAS) ranging from 0 (no impact on quality of life) to 100 (worst possible impact). Thus, the total score ranged from 0 to 2100 points. The score was reported as a percentage of normal by subtracting the total score from 2100, dividing by 2100, and multiplying by 100. Total final WORC percentage scores ranged from 0%, the lowest functional status level, to 100%, the highest functional status level.
  Change from baseline in the WORC percentage total score was assessed at Week 24. A positive change from baseline indicated an improvement.
Time Frame: Baseline, Week 24
Population: FAS: all patients to whom study/reference treatment was assigned by randomization.
  Only participants with both a baseline and a Week 24 assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 28 | 28
Score on a Scale | 55.7 (28.1) | 46.8 (26.9)

2. Secondary Outcome: Change From Baseline in the WORC Percentage Sub-scores at Week 24
Description: The WORC Index consisted of 21 items divided into 5 Domains: Physical Symptoms (6 items), Sport/Recreation (4 items), Work Function (4 items), Lifestyle Function (4 items) and Emotional Function (3 items). Each of the 21 items in the WORC was rated using a VAS ranging from 0 (no impact on quality of life) to 100 (worst possible impact).
  Each subdomain score was calculated as a percentage of normal function, ranging from 0% (worst condition) to 100% (best condition).
  Change from baseline in the WORC Index percentage sub-domain score was assessed at Week 24. A positive change from baseline indicated an improvement
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 28 | 28
Score on a Scale
  Physical symptom score | 48.8 (31.2) | 40.0 (25.0)
  Sports and recreation | 51.8 (30.9) | 44.0 (30.6)
  Work | 59.7 (32.0) | 49.9 (30.5)
  Lifestyle | 59.5 (27.3) | 52.9 (26.4)
  Emotional function | 64.2 (23.6) | 54.3 (31.5)

3. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity Score at Week 24
Description: The participant's global assessment of disease activity was performed using 100 mm VAS ranging from 0="no activity" to 100= "most active", after the question " Please indicate with a vertical mark ( | ) through the horizontal line the global activity of your disease in the last 24 hours".
  Change from baseline in the participant's global assessment of disease activity score was assessed at Week 24. A negative change from baseline indicated improvement
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 26 | 25
Score on a scale | -46.4 (36.6) | -18.5 (37.2)

4. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36v2) Score at Week 24
Description: The SF-36 Health Survey was a validated questionnaire assessing health-related quality of life. Participants completed the survey throughout the study, reflecting their health status over the previous 4 weeks. It consisted of eight subscales that were scored individually; and two overall summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Component summary scores (PCS and MCS) were derived from weighted combinations of the eight subscales. Each domain and component summary score ranged from 0 to 100, with higher scores indicating better quality of life.
  Change from baseline to Week 24 in all subscale and summary scores was assessed, where a positive change indicated improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 26 | 25
Score on a Scale
  Physical component summary | 9.4 (9.1) | 9.7 (7.9)
  Mental component summary | 8.0 (10.7) | 6.3 (11.9)
  General health | 3.0 (8.5) | 3.9 (10.6)
  Vitality | 8.3 (9.9) | 7.7 (11.0)
  Social functioning | 8.3 (10.1) | 8.2 (10.9)
  Role emotional | 11.5 (13.1) | 5.8 (14.5)
  Mental health | 7.6 (10.0) | 9.1 (10.9)
  Physical function | 8.8 (9.5) | 8.6 (6.4)
  Role-physical | 9.9 (10.3) | 9.3 (10.9)
  Bodily pain | 16.2 (10.2) | 15.1 (9.2)

5. Secondary Outcome: Change From Baseline in Quick Disability of the Arm, Shoulder and Hand (DASH) Questionnaire Score at Week 24
Description: The QuickDASH was an abbreviated form of the DASH. The QuickDASH Index was self-administered and used 11 items to measure physical function and symptoms in participants with any or multiple musculoskeletal disorders of the upper limb. It had a recall period of 1 week. Each item of the QuickDASH had five response options. The raw score was calculated as the sum of responses, converted to an average, and rescaled to a total score ranging from 0 (no disability) to 100 (most severe disability) Change from baseline to Week 24 was assessed. A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 26 | 25
Score on a Scale | -34.1 (23.7) | -33.5 (24.6)

6. Secondary Outcome: Change From Baseline in the Numeric Rating Scale (NRS) Pain Score at Week 24
Description: The score for pain was assessed by using an 11-point NRS ranging from 0 "no pain at all" to 10 "worst possible pain", after the question "On a numeric scale of 0-10 where would you rate your pain at this time".
  Change from baseline to Wek 24 was assessed. A negative change from baseline indicated improvement
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 26 | 25
Score on a Scale | -4.5 (2.8) | -4.6 (2.4)

7. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions- 5 Levels (EQ-5D-5L) at Week 24- Total Score
Description: The EQ-5D-5L was a standardized instrument used to evaluate patients' overall health-related quality of life (QoL). It consisted of two components: the descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system assessed five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension was rated on five levels, from 1 (no problems) to 5 (extreme problems). These ratings were combined to generate a composite health index, which could be converted into a single summary health utility score using published value sets. Total scores ranged from 0 to 1, with lower scores indicating greater health impairment.
  Changes in total scores from baseline to Week 24 were analyzed, with positive changes indicating improvement in health-related quality of life.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 26 | 25
Score on a Scale | 0.265 (0.226) | 0.342 (0.228)

8. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions- 5 Levels (EQ-5D-5L) at Week 24- EQ VAS
Description: The EQ-5D-5L was a standardized instrument used to evaluate patients' overall health-related quality of life (QoL). It consisted of two components: the descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ VAS captured the respondent's self-rated health on a vertical scale ranging from 0 (worst imaginable health) to 100 (best imaginable health).
  Changes in EQ VAS scores from baseline to Week 24 were analyzed, with positive changes indicating improvement in health-related quality of life.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 26 | 25
Score on a Scale | 18.3 (36.5) | 23.8 (27.3)

ADVERSE EVENTS:
Time Frame: From start of treatment to end of study, assessed up to approximately 24 weeks
Description: The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Groups:
- Secukinumab; Placebo: AEs from start of treatment to 84 days after the last dose of study treatment, assessed up to approximately 24 weeks
Arm/Group | Secukinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/30 | 3/32
Other Adverse Events (participants affected / at risk) | 22/30 | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=30) | Placebo (N=32)
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Vaginal cuff dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Occipital lobe stroke (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Paradoxical embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=30) | Placebo (N=32)
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders and administration site conditions) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 3
COVID-19 (Infections and infestations) | 4 | 3
Gastrointestinal infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 5 | 7
Oral herpes (Infections and infestations) | 2 | 2
Respiratory tract infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 8 | 6
Depression (Psychiatric disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT05569174/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT05569174/SAP_001.pdf